CLINICAL TRIAL: NCT05240183
Title: Viral Dynamics of the SARS-CoV-2 Omicron Variant in Paediatric Patients
Brief Title: Viral Dynamics of Omicron in Children
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Michelle Science, Infectious Disease Physician, The Hospital for Sick Children
Other Study IDs: 1000079263
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: SARS-CoV2 Infection, COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Daily SARS-CoV-2 PCR Testing for 10 days — Each participant will undergo daily SARS-CoV-2 PCR testing to assess viral dynamics

SUMMARY:
SARS-CoV-2 transmission is dependent on multiple factors, which may be related to either host-virus interaction or the environment. While there have been several studies evaluation viral dynamics and transmission risk in adults, there is limited pediatric data available. The objective of this study is to characterize the period of communicability for children less than 19 years of age with SARS-CoV-2 infection with the Omicron variant.

DETAILED DESCRIPTION:
The goal of our study is to assess the viral dynamics of SARS-CoV-2 infection in children < 19 years with acute infection to inform public health practice.

Specific Aims:

1. Describe the kinetics of SARS-CoV-2 viral load in children with acute SARS-CoV-2 infection
2. Assess the impact of various host factors on viral dynamics, including age (<1 year, 1-4 years, 5-11 years, 12-18 years), symptoms, clinical severity (hospitalization vs. outpatient), comorbidities (immunocompromised vs. not immunocompromised), vaccination (none, 1 dose, 2 doses)
3. Estimate the time point at which children are less likely to be infectious
4. Assess the sensitivity of self-collected rapid antigen testing (RAT) in children, compared to PCR (e.g. assess RAT test performance in children)

ELIGIBILITY:
To be included in the study, the participant must be:

1. Less than 19 years of age
2. Have a positive molecular or rapid antigen test in the previous 48 hours
3. If symptomatic, onset of any COVID-19 symptom within last 72 hours.
4. If asymptomatic, evidence to support acute infection (e.g. negative PCR in the last 5 days, known household exposure where index case is clear)
5. Able to collect daily samples

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children less than 19 years of age with acute SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 Viral Load | 10 days
  We will use prospective longitudinal quantitative reverse transcription PCR testing to measure the viral RNA trajectories for individuals in the study.

SECONDARY OUTCOMES:
Rapid antigen test sensitivity | 10 days
  We will describe the RAT positivity on Days 1 to 10 and evaluate the performance of RAT compared to PCR

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Science M, Orkin J, Maguire B, Bitnun A, Bourns L, Corbeil A, Johnstone J, Macdonald L, Schwartz KL, Bruce Barrett C, Reinprecht J, Heisey A, Nasso S, Juni P, Campigotto A. Viral Dynamics of the SARS-CoV-2 Omicron Variant in Pediatric Patients: A Prospective Cohort Study. Clin Infect Dis. 2024 Jun 14;78(6):1506-1513. doi: 10.1093/cid/ciad740. PMID 38084906